CLINICAL TRIAL: NCT05305027
Title: Single-centre Retrospective Study on the Predictive Value of Sequential Early βHCG Measurements in IVF Pregnancies.
Brief Title: Predictive Value of Sequential βHCG in IVF Pregnancy
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Research Administration Manager and Head of Clinical Trial Office Humanitas Clinical and Research Center, Istituto Clinico Humanitas
Other Study IDs: 21012021
Record Dates: First submitted 2022-02-03; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Early

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IVF patients: first serum βHCG: IVF patients who undergo βHCG after fresh or frozen embryo transfer
  Interventions: Behavioral: Prompt diagnois pregnancy outcome

INTERVENTIONS:
Behavioral: Prompt diagnois pregnancy outcome

SUMMARY:
Early diagnosis of pregnancy with its localization and evolution has always been one of the major objectives of gynecology and obstetrics, even more so in Artificial Reproductive Technology (ART) centers.

The pivotal test is the βHCG assay. Various protocols have been proposed over the years, including single assessment and serial assays.

Several studies in the past years have tried to define a cut-off predictive of a successful pregnancy.

Abnormal levels of βHCG are associated with biochemical pregnancies, non-viable pregnancies and ectopic pregnancies (EP). The efficacy of a single serum βHCG test to predict EP is low and a significant amount of time and resources are spent diagnosing it.

In recent studies, better sensitivity was obtained from the ratio of two successive time points of βHCG concentration, with better specificity instead from regression models. These proposed models however lack validation and require further improvement.

DETAILED DESCRIPTION:
Fertility clinics follow different protocols for the measurement of βHCG. Typically the initial serum measurement is performed 10-12 days after blastocyst transfer or 12-14 days after transfer at cleavage stage. Often a second serum measurement of hCG is performed at 48h since an increase of at least 50% is known to be a good predictor of ongoing pregnancy.

The doubling time was first described in natural pregnancies where the rate of βHCG rise was reported to be at least 53% in two days, with a median of 50% increase at day 1 and 124% at day 2. Following the first detection and rise of serum βHCG, it is possible to predict earlier than with transvaginal ultrasound non-viable pregnancies, ectopic pregnancies, biochemical pregnancies and spontaneous abortion or reassure the couple when these values are representative of an ongoing pregnancy (OP). Conversely, however, many studies have found different thresholds of βHCG to be representative of OP, with many women under the cut-off value ending up having a normal pregnancy.

The variability within the threshold expresses the need for a better biological marker or cut-off value. Implementing patient characteristics in a model to redefine and personalize the cut-off is necessary to improve pregnancy detection and management.

ELIGIBILITY:
All women that underwent IVF cycles (including fresh and thawed embryo transfers) between January 2011 and December 2020.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include retrospectively all patients that underwent IVF cycles (including fresh and thawed embryo transfers) between January 2011 and December 2020 at a Third level University-affiliated center, Humanitas Fertility Center in (Rozzano, MI).
  The internal database (Art-it) will be used to retrieve data on age, body mass index (BMI), baseline sex hormone levels, main causes of infertility, endometrial thickness, details of stimulation protocols, date of insemination, date of embryo transfer, number of embryos transferred, date of βHCG examination, serum concentrations of βHCG, fertilization results, pregnancy types (EP, biochemical pregnancy, intrauterine)
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Live birth incidence per serum βHCG value | 1 year
  Compare the incidence of Live Birth according to serum βHCG (IU/L) measurement in all patients undergoing ART procedures.

SECONDARY OUTCOMES:
Comparison of live birth incidence with serum βHCG confounders | 1 year
  Comparison of live birth incidence according to possible risk factors for serum βHCG (IU/L) measurements, among patients undergoing ART procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Emanuele Levi Setti, MD, Study Director — Istituto Clinico Humanitas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seeber BE, Sammel MD, Guo W, Zhou L, Hummel A, Barnhart KT. Application of redefined human chorionic gonadotropin curves for the diagnosis of women at risk for ectopic pregnancy. Fertil Steril. 2006 Aug;86(2):454-9. doi: 10.1016/j.fertnstert.2005.12.056. Epub 2006 Jun 6. PMID 16753158
- [Result] Wang Z, Gao Y, Zhang D, Li Y, Luo L, Xu Y. Predictive value of serum beta-human chorionic gonadotropin for early pregnancy outcomes. Arch Gynecol Obstet. 2020 Jan;301(1):295-302. doi: 10.1007/s00404-019-05388-2. Epub 2019 Nov 22. PMID 31758302